CLINICAL TRIAL: NCT00415324
Title: A Phase 1 Study of Halichondrin B Analog (E7389) in Combination With Cisplatin in Advanced Solid Tumors
Brief Title: Eribulin Mesylate and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00168; NCI-2009-00168 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-55; CDR0000518290; PHI-55 (Other: City of Hope Medical Center); 7427 (Other: CTEP); U01CA062505 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — eribulin; Cisplatin

ARMS (1):
- Arm 1 (Experimental): Patients receive eribulin mesylate IV over 5 minutes on days 1, 8, and 15 and cisplatin IV over 30-60 minutes on day 1.
  Interventions: Drug: eribulin mesylate; Drug: cisplatin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: laboratory biomarker analysis — correlative study
Other: pharmacological study — correlative study
  Other Names: pharmacological studies

SUMMARY:
This trial is studying the side effects and best dose of eribulin mesylate and cisplatin in treating patients with advanced solid tumors.Drugs used in chemotherapy, such as eribulin mesylate and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
Primary Objectives:

I. To determine the maximum tolerated dose of E7389 and cisplatin in patients with advanced solid tumors.

II. To determine the safety and toxicity of this regimen in these patients. III. To determine the pharmacokinetics of this regimen in these patients.

Outline: This is a multicenter, dose-escalation study. Patients receive eribulin mesylate IV over 5 minutes on days 1, 8, and 15 and cisplatin IV over 30-60 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant solid tumor
* Advanced disease, meeting both of the following criteria: Metastatic or unresectable disease and standard curative or palliative measures do not exist or are no longer effective.
* No known active brain metastases
* Life expectancy > 3 months
* ECOG performance status 0-2
* Bilirubin normal
* No uncontrolled intercurrent illness including, but not limited to, any of the following: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness or social situation that would limit study compliance.
* Negative pregnancy test
* Fertile patients must use effective contraception
* Recovered from prior therapy
* No prior chemotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C).
* No prior targeted therapy within the past 4 weeks
* No prior immunotherapy within the past 4 weeks
* No prior radiotherapy within the past 4 weeks.
* No more than 2 prior chemotherapy regimens for advanced solid tumors.
* No other concurrent investigational agents. Bisphosphonate therapy (e.g., pamidronate or zolendronate) is not considered investigational therapy.
* No concurrent antiretroviral therapy for HIV-positive patients.
* No other concurrent anticancer agents or therapies.
* Tumor has spread to other parts of the body or cannot be removed by surgery.
* More than 4 weeks since chemotherapy, biological therapy, or radiation therapy.
* No more than two previous chemotherapy regimens for advanced solid tumor.
* WBC >= 3,000/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine clearance >= 60 mL/min
* Absolute neutrophil count >= 1,500/mm³
* AST and ALT =< 2.5 times upper limit of normal
* No prior cumulative cisplatin dose > 300 mg/m^2
* No preexisting neuropathy <= grade 2
* Not pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-12; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicity graded according to the NCI CTCAE version 4.0 | 28 days

SECONDARY OUTCOMES:
Survival | From first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 8 weeks
  Summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol.
Time to failure | Up to 8 weeks
  Summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Koczywas, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - City of Hope, Duarte, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - University of California at Davis Cancer Center, Sacramento, California